CLINICAL TRIAL: NCT06518577
Title: Measuring Immunity Against Circulating Influenza Viruses: Randomized Immunogenicity Study Among US Adults Aged 18-64 Years Comparing Two Approved Influenza Vaccines
Brief Title: Immunogenicity of Influenza Vaccinations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Arizona State University (Other); University Hospitals Cleveland Medical Center (Other); University of Pittsburgh (Other); Washington University School of Medicine (Other); VA Medical Center-Cleveland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00115120
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Influenza
Keywords: Influenza; Immunogenicity
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; FluBlok

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Flucelvax (ccIIV4) (Experimental): Participants will receive Flucelvax (ccIIV4) at Visit 1.
  Interventions: Biological: Flucelvax (ccIIV4)
- Flublok (RIV) or Fluzone (IIV) (Experimental): Participants will receive Flublok (RIV) or Fluzone (IIV) at Visit 1.
  Interventions: Biological: Flublok (RIV) or Fluzone (IIV)

INTERVENTIONS:
Biological: Flucelvax (ccIIV4) — Participants will receive Flucelvax (ccIIV4)
  Arms: Flucelvax (ccIIV4)
Biological: Flublok (RIV) or Fluzone (IIV) — Participants will receive Flublok (RIV) or Fluzone (IIV)
  Arms: Flublok (RIV) or Fluzone (IIV)

SUMMARY:
This study is a randomized immunogenicity study in an enrolled cohort with active surveillance for influenza-like illness (ILI). During this study, participants will be randomly assigned to receive an approved cell culture-based influenza vaccine (Flucelvax) versus a licensed comparator influenza vaccine (Flublok or Fluzone). Blood samples from participants will be collected for measurement of biomarkers of immune response at baseline (visit 1; day 1), post-vaccination (visit 2; day 29), and post-season (visit 3; day 181). Participants will be asked if they wish to also provide saliva specimens at baseline (visit 1; day 1), post-vaccination (visit 2; day 29), and post-season (visit 3; day 181). Serum and peripheral blood mononuclear cells (PBMC) and plasma samples will be isolated from whole blood and tested for biomarkers of vaccine immunogenicity, and duration of antibody responses.

Participants will receive electronic surveys via email or text message weekly asking about changes in health status and new ILI symptoms; those reporting illness may be asked to provide a respiratory swab for laboratory testing for influenza and other respiratory viruses and up to 2 additional blood draws (acute [<10 days after symptom onset] and convalescent [28 days after acute visit if lab-confirmed positive for influenza]).

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18-64 years that have not received the current season's influenza vaccine
2. English literate
3. Email or text message capability for weekly follow-up
4. Intention of receiving influenza vaccine based on ACIP-CDC guidelines
5. Willing to provide written/electronic informed consent
6. Intention of being available for entire study period and able to complete all relevant study procedures, including follow-up phone calls and clinic visits

Exclusion Criteria:

1. Receipt of the current season's influenza vaccine (receipt after July 1, 2024)
2. History of severe allergic reaction after a previous dose of any influenza vaccine or to an influenza vaccine component
3. Receipt of any licensed or investigational live vaccine within 6 weeks or non-live vaccine within 2 weeks prior to enrollment in this study or planning receipt of any vaccines between visits 1 and 2 of the study (approximately within 4 weeks after the receipt of study-administered vaccine)
4. History of Guillain-Barré syndrome
5. Currently pregnant, planning to become pregnant within the first three months of the study per participant self-report
6. Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
7. Any condition which, in the opinion of the investigators, may pose a health risk to the participant or interfere with the evaluation of the study objectives

Temporary Delay Criteria (Visit 1)

1. History of febrile illness (> 100.0°F or 37.8°C) within the past 72 hours prior to vaccine administration

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 605 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Participants with a seroprotective HAI titer (≥1:40) | Baseline, Day 29
  The number (percent) of participants with a seroprotective HAI titer (≥1:40) for each influenza vaccine antigen
The geometric mean titer (GMT) of HAI antibody | Baseline, Day 29
  The geometric mean titer (GMT) of HAI antibody for each influenza vaccine antigen
Number of participants demonstrating seroconversion from baseline | Day 29
  The number (percent) of participants in each vaccination group demonstrating seroconversion from Baseline at Day 29 (a titer ≥1:40 at Day 29 if the baseline titer is <1:10 or a four-fold rise in titer at Day 29 if the baseline titer is >1:10) as assessed by HAI titer for each vaccine antigen
Geometric mean fold rise (GMFR) in HAI titer from baseline | Day 29
  The geometric mean fold rise (GMFR) in HAI titer from Baseline to Day 29 across HAI titers for each influenza vaccine antigen

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel B Walter, MD, MPH, Principal Investigator — Duke University
Locations (7):
- United States (7):
  - Valleywise Health Comprehensive Health Center, Phoenix, Arizona
  - ASU Biodesign Institute, Tempe, Arizona
  - Centers for Disease Control and Prevention, Atlanta, Georgia
  - Washington University IDCRU, St Louis, Missouri
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - VA Northeast Ohio Healthcare System (VANEOHS), Cleveland, Ohio
  - Department of Family Medicine, University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-09-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT06518577/ICF_000.pdf